CLINICAL TRIAL: NCT04591587
Title: Corneal Lenticule Implantation in Keratoconus Disease With Relex Smile Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Faruk Semiz (Other)
Responsible Party: Sponsor-Investigator, Dr. Faruk Semiz, Principal Doctor, Eye Hospital Pristina Kosovo
Organization: Eye Hospital Pristina Kosovo (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EyeHPristina
Record Dates: First submitted 2020-06-15; First posted 2020-10-19 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Keratoconus
Keywords: Keratoconus; Small Incision; Fresh Lenticule; Stromal Implantation; Stromal Stem Cells; Smile Surgery
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Intervention Model Description: Both models participated in this study. Model ages were from 20 up to 45
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smile Group (Active Comparator): Twenty patients (20) underwent SMILE surgery (first group)
  Interventions: Procedure: Lenticule Implantation in Keratoconus Disease with RELEX Smile Surgery
- Lenticule Group (Active Comparator): Twenty patients (20) underwent lenticule implantation (second group)
  Interventions: Procedure: Lenticule Implantation in Keratoconus Disease with RELEX Smile Surgery

INTERVENTIONS:
Procedure: Lenticule Implantation in Keratoconus Disease with RELEX Smile Surgery — Lenticule Implantation in Keratoconus Disease with RELEX Smile Surgery using VisuMax Femtosecond laser- Smile module surgery with primary objective to increase central corneal thickness and secondary objective to improve visual acuity and reduces K-values

SUMMARY:
CORNEAL LENTICULE IMPLANTATION IN KERATOCONUS DISEASE WITH RELEX SMILE SURGERY

DETAILED DESCRIPTION:
Purpose:

The purpose of our study is to investigate the feasibility and effect of fresh lenticule implantation as allogenic graft that will be taken from myopic patients, in order to implant in patients with keratocouns disease using VisuMax Femtosecond laser - Smile module surgery which primary objective in to increase central corneal thickness and secondary objective is to improve visual acuity and reducing K-values.

Methods:

All the patients were clinically diagnosed with progressive keratoconus. Twenty (20) patients underwent SMILE surgery (first group), and twenty (20) patients underwent lenticule implantation (second group). Visual acuity, corneal topography, electron microscop,anterior segment optical coherence tomography, were analyzed.

Outcome:

Central corneal thickness were improved at the same day of surgery and vision started to improve at first week postoperatively in the second group (lenticule implant group). Corneal topography showed a statistically significant decrease in the anterior K1 and K2. All the grafts from both groups were clearly visible by anterior segment optical coherence tomography observation and electron microscope. The central corneal thickness was stable during the 6-month study period. No complications were observed during short term follow-up.

Opinion:

In our opinion, the present study may suggest that this procedure, using fresh lenticule with stromal stem cells and live keratocites is safe, reliable, and effectively increases corneal thickness and improves visual acuity with no adverse effects, which may provide new avenues in the treatment of corneal ectasia.

Key Words:

keratoconus,small incision,fresh lenticule, stromal implantation,stromal stem cells, Smile surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed with progressive keratoconus

Exclusion Criteria:

* Active anterior segment pathologic features, Corneal thickness over 420, Previous corneal or anterior segment surgery

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Increase of corneal thickness at patients Lenticule group | 12 months
  Increase of corneal central thickness using fresh lenticule with stromal stem cells and live keratocytes

SECONDARY OUTCOMES:
Improvement of visual acuity at patients Lenticule group | 12 months
  Increase of visual acuity using fresh lenticule, decrease of astigmatism and increase of corneal thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital Pristina, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-06-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT04591587/ICF_000.pdf